CLINICAL TRIAL: NCT07294235
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single/Multiple-dose Study to Evaluate the Tolerability, Safety and Pharmacokinetics of BGM1812 in Healthy and Non-diabetic Overweight or Obese Chinese Participants
Brief Title: A Study of BGM1812 Injection in Healthy and Non-diabetic Overweight or Obese Chinese Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Collaborators: BrightGene Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGM1812-CPK-101
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BGM1812(Part A) (Experimental): Single ascending doses of BGM1812 administered subcutaneously (SC)
  Interventions: Drug: BGM1812
- Placebo (Part A) (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- BGM1812 (Part B) (Experimental): Multiple ascending doses of BGM1812 administered SC.
  Interventions: Drug: BGM1812
- Placebo (Part B) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGM1812 — AdministeredSC
  Arms: BGM1812(Part A)
Drug: Placebo — Administered SC
  Arms: Placebo (Part A)
Drug: BGM1812 — Administered SC
  Arms: BGM1812 (Part B)
Drug: Placebo — Administered SC
  Arms: Placebo (Part B)

SUMMARY:
The purpose of this study is to evaluate the tolerability , safety and pharmacodynamics of BGM1812 administered subcutaneously in healthy and non-diabetic overweight or obese Chinese participants, and to investigate the pharmacokinetic profile of BGM1812 in the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years (inclusive) at the time of screening , healthy and non-diabetic overweight or obese subjects , both male and female;
* Healthy subjects , male weight ≥ 50 kg, female weight ≥ 45 kg, and body mass index (BMI): 20.0 kg/m² ≤ BMI < 24 kg/m²（BMI = weight/height²）;
* Obese individuals: BMI ≥ 28.0 kg/m², or overweight individuals: 24.0 kg/m² ≤ BMI < 28.0 kg/m²;
* (Medical Inquiry) Have a stable body weight (<5% self-reported change during the previous 12 weeks) before screening.
* Have no history of mental disorders, be able to communicate smoothly with Investigator, Capable of understanding the written informed consent document; willingly provides valid, signed written informed consent; willing and able to comply with the schedule, requirements and restrictions of the study.
* Male subjects with female partners of reproductive potential must agree to practice abstinence or to use a condom (male subject) plus an additional medically acceptable form of contraception (female partner) for the duration of the study and for at least 3 months after dosing; must also agree to refrain from sperm donation for at least 3 months post dose.

Exclusion Criteria:

* Those with a history of severe drug allergies (especially those with known or suspected allergies to related compounds of BGM1812), or complicated with severe specific allergic diseases/history, or with a severe allergic constitution.
* Subjects with positive results for HBsAg, anti-HCV, anti-HIV or anti-TP during the screening period.
* 12-lead ECG shows ventricular heart rate < 50 beats/min or > 100 beats/min at screening/baseline, second or third degree atrioventricular block, long QT syndrome, QTcF> 470ms for women or > 450ms for men, pre-excitation syndrome or other significant arrhythmias.
* Used illegal drugs within 6 months prior to screening, or substance abuse within 12 months prior to screening.
* Participated in drug or medical device clinical trials and treated with Study Drug (excluding placebo) or medical device intervention within 12 weeks before screening.
* Participants who have received any vaccine within 2 weeks prior to screening, or plan to receive a vaccine during the trial.
* Female participants who are pregnant or lactating, or those with a positive pregnancy test result during the screening period.
* Positive urine drug test or alcohol serum test result at screening or at baseline.
* Has any other conditions or disorders deemed unsuitable for including in the study, in the opinion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Events (AEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator | Baseline to Study Completion (Up to 6-9weeks)
  Number of participants with AEs and SAEs will be assessed with reference to CTCAE V5.0

SECONDARY OUTCOMES:
Pharmacokinetic (PK): Maximum Concentration (Cmax) of BGM1812 | Baseline to Study Completion (Up to 6-9weeks)
  PK Cmax of BGM1812
PK: Area Under the Concentration Versus Time Curve (AUC) of BGM1812 | Baseline to Study Completion (Up to 6-9weeks)
  PK:AUC of BGM1812
Pharmacodynamics (PD): Fasting Blood Glucose of BGM1812 | Baseline to Study Completion (Up to 6-9weeks)
  PD: Changes in fasting blood glucosebefore and after administration, and differences in the amount of change among different dose groups
PD:C-Peptide of BGM1812 | Baseline to Study Completion (Up to 6-9weeks)
  PD: Changes in C-peptide before and after administration, and differences in the amount of change among different dose groups
PD: Insulin of BGM1812 | Baseline to Study Completion (Up to 6-9weeks)
  PD: Changes in insulin before and after administration, and differences in the amount of change among different dose groups
PD: Body Weight of BGM1812 | Baseline to Study Completion (Up to 6-9weeks)
  PD: Changes in body weight before and after administration, and differences in the amount of change among different dose groupsPD: Changes in body weight before and after administration, and differences in the amount of change among different dose groups
PD: Waist Circumference of BGM1812 | Baseline to Study Completion (Up to 6-9weeks)
  PD: Changes in waist circumference before and after administration, and differences in the amount of change among different dose groups
Immunogenicity Endpoints | Baseline to Study Completion (Up to 6-9weeks)
  Detect the anti-drug antibodies (ADA) of the study drug and their titers; if the ADA is positive, neutralizing antibodies (NAb) will be further detected.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Yunnan University of Chinese Medicine, Kunming, Yunnan, China